CLINICAL TRIAL: NCT02334605
Title: Comparison of Cold Dry Air Exposure, Hyperosmolar Sponge and Capsaicin Nasal Spray for Objective Evaluation of Nasal Hyperreactivity
Brief Title: Comparison of Cold Dry Air Exposure, Discs and Capsaicin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CDAvsDiscsvsCap
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Nasal Hyper Reactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cold dry air (Other): Patients will be asked to acclimatize to room temperature for 20 minutes prior to exposure to cold dry air.
  Through a nasal cannula, compressed dry air for medical use will be delivered for 15 minutes (25L/minute). Patients will be instructed to breathe through the nose only. The temperature of the air reaching the nose will be approximately -10°C and the relative humidity less than 10-15%.
  Interventions: Other: cold dry air
- hyperosmolar discs (Other): A small paper disc (5-6mm of diameter) previously loaded with 50µl NaCl 5,13M will be applied on the right nasal septum for 1 minute and then be discarded.
  Interventions: Device: hyperosmolar discs
- capsaisin nasal spray (Other): one puff of a nasal spray with a solution of capsaicin 0,0001mM will be sprayed in each nostril of the subject and subjects will be asked to score visual analogue scale for irritation of the nasal mucosa immediately after the adminitration.
  Interventions: Device: capsaicin nasal spray

INTERVENTIONS:
Other: cold dry air — Patients will be asked to acclimatize to room temperature for 20 minutes prior to exposure to cold dry air.
  Through a nasal cannula, compressed dry air for medical use will be delivered for 15 minutes (25L/minute). Patients will be instructed to breathe through the nose only. The temperature of the air reaching the nose will be approximately -10°C and the relative humidity less than 10-15%.
  Arms: cold dry air
Device: hyperosmolar discs — A small paper disc (5-6mm of diameter) previously loaded with 50µl NaCl 5,13M will be applied on the right nasal septum for 1 minute and then be discarded.
  Arms: hyperosmolar discs
Device: capsaicin nasal spray — 1 puff of a nasal spray with a solution of capsaicin 0,0001mM will be sprayed in each nostril of the subject and subjects will be asked to score visual analogue scale for irritation of the nasal mucosa immediately after the adminitration.
  Arms: capsaisin nasal spray

SUMMARY:
Nasal hyper reactivity is defined as an increased sensitivity of the nasal mucosa to stimuli such as temperature changes, changes in humidity, emotional stress, physical activity, smoke and/or other scents and gives often rise to nasal symptoms such as rhinorrhea, nasal obstruction and/or sneezing.

nasal hyper reactivity is a clinical feature of rhinitis and rhinosinusitis, affecting more than 20% of the total Western population.

Cold, dry air exposure has been shown to be a reliable method for diagnosis of nasal hyperreactivity. The new, shorter protocol for cold dry air provocation that recently has been validated as a useful diagnostic tool to evaluate nasal hyperreactivity with high specificity and sensitivity, is already a major step forward but still rather time-consuming and not always very practical in use.

A hyperosmolar saline solution loaded on a small nasal sponge as described earlier has also been reported as being an effective means of evaluation of nasal hyperreactivity. In addition, capsaicin nasal spray has also been reported as being an elegant tool for the evaluation of the response of TRP channels on the nasal mucosa.

So far, we lack data on the comparison between the 3 different diagnostic tools for the evaluation of nasal hyperreactivity in rhinitis.

ELIGIBILITY:
Inclusion Criteria:

DM AR patients with at least two nasal complaints rhinorrhea, nasal obstruction, itch or sneezing.

* HDM AR patients with a total nasal symptoms score (TNS) of 5 or more on a visual analogue scale (VAS).
* HDM AR patients with positive skin prick test (Hal reagents) for house dust mite and/or IgE in blood. *
* IR patients with at least two nasal complaints rhinorrhea, nasal obstruction, itch or sneezing.
* IR patients with a total nasal symptoms score (TNS) of 5 or more on a visual analogue scale (VAS).
* HC with no rhinological complaints during the previous three months with negative skin prick test (Hal reagents) for the 18 most frequent aeroallergens in Belgium. *
* Age > 18 and < 65 years.
* Written informed consent.
* Willingness to adhere to the planned visits.

Exclusion Criteria:

* Individuals with structural abnormalities: nasal polyps, severe septal deviation (septum reaching concha inferior or lateral nasal wall), septal perforation, hypertrophy of the inferior turbinates.

  * Individuals with local allergic rhinitis (LAR) or entopy.
  * Systemic steroid treatment less than 4 weeks before the inclusion in the study, nasal steroid spray less than 4 weeks before the inclusion, oral leukotriene antagonists or long-acting antihistamines less than 2 weeks before the inclusion.
  * Inability of the person to stop taking medication affecting nasal function like ß-blockers.
  * History of prolonged use or abuse of decongestant nasal spray like xylometazoline spray and/or use or abuse of decongestive oral medication.
  * Evidence of infectious rhinitis/rhinosinusitis or common cold within 4 weeks prior to inclusion.
  * Any disorder of which might compromise the ability of a patient to give truly informed consent for participation in this study.
  * Enrollment in other investigational drug trial(s) or receiving other investigational agent(s) for any other medical condition.
  * Smoking or occupational exposure to irritants (like hypochlorite, persulfates, isocyanates).
  * Nasal malignancies or severe comorbidity like granulomatosis or vasculitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in peak nasal inflamatorry flow | baseline, 5 minutes

SECONDARY OUTCOMES:
change of nasal symptom visual analogue scale | baseline, 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: peter hellings, Prof Dr, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven ENT, Leuven, Vlaams Brabant, Belgium